CLINICAL TRIAL: NCT05705388
Title: Comparison of Efficacy and Safety of POSE 2.0 Procedure Compared to GLP-1 Agonist in a Cohort of Patients for Management of Obesity: a Single-center Randomized Crossover-controlled Trial
Brief Title: POSE2.0 With GLP-1 Agonist for Obesity Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Emirates Health Services (EHS) (Other Government)
Responsible Party: Principal Investigator, Mariam Salem Alkhatry, Head of Endoscopy, Division of Gastroenterology, Ibrahim Bin Hamad Obaidullah Hospital, Ras Al Khaimah, United Arab Emirates, Emirates Health Services (EHS)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UAE_V1
Record Dates: First submitted 2023-01-09; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: 6 months of liraglutide (titrated to 3mg daily or maximal tolerated dose) or 6 months of POSE 2.0 with both groups receiving combination of both therapies for 6 months if they did not reach a BMI less than 30kg/m2 at the time of cross-over at 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- POSE2.0 Procedure (Active Comparator): The POSE2.0 is a per-oral endoscopic gastroplasty procedure performed by the USGI Medical Incisionless Operating Platform (USGI Medical, San Clemente, CA) to deploy preloaded snowshoe suture anchors, and cinch create gastric endoscopic plications. In the POSE2.0 procedure a series of 15-20 pairs of snowshoes anchors are deployed along the greater curvature of the stomach from the proximal antrum to the proximal gastric body along narrowing the anteroposterior diameter of the stomach and decreasing its vertical length to improve satiety and satiation for weight loss. This device is registered and approved for obesity management in the United Arab Emirates, where the study is performed.
  Interventions: Device: POSE2.0 Endoscopic Gastric Remodeling; Drug: Liraglutide injection
- Liraglutide (Active Comparator): Liraglutide is a GLP-1 agonists approved for the management of obesity. In the study, it will be Initiated at 0.6 mg subcutaneously daily for 1 week; increase by 0.6 mg/day in weekly intervals until a dose of 3 mg/day achieved. If patients do not tolerate an increased dose during dose escalation, dose escalation will be delayed for an additional week. The patient will continue at the maximal tolerated does up to 3mg per day. If the patient has not lost at least 4% of baseline body weight at 16 weeks from medication initiation, the medication will be discontinued.
  Interventions: Device: POSE2.0 Endoscopic Gastric Remodeling; Drug: Liraglutide injection

INTERVENTIONS:
Device: POSE2.0 Endoscopic Gastric Remodeling — The POSE2.0 is a per-oral endoscopic gastroplasty procedure performed by the USGI Medical Incisionless Operating Platform (USGI Medical, San Clemente, CA) to deploy preloaded snowshoe suture anchors, and cinch create gastric endoscopic plications. In the POSE2.0 procedure a series of 15-20 pairs of snowshoes anchors are deployed along the greater curvature of the stomach from the proximal antrum to the proximal gastric body along narrowing the anteroposterior diameter of the stomach and decreasing its vertical length to improve satiety and satiation for weight loss. This device is registered and approved for obesity management in the United Arab Emirates, where the study is performed.
Drug: Liraglutide injection — Liraglutide is a GLP-1 agonists approved for the management of obesity. In the study, it will be Initiated at 0.6 mg subcutaneously daily for 1 week; increase by 0.6 mg/day in weekly intervals until a dose of 3 mg/day achieved. If patients do not tolerate an increased dose during dose escalation, dose escalation will be delayed for an additional week. The patient will continue at the maximal tolerated does up to 3mg per day. If the patient has not lost at least 4% of baseline body weight at 16 weeks from medication initiation, the medication will be discontinued.

SUMMARY:
Determine the effect on weight loss and obesity-related comorbidities in patients receiving the POSE 2.0 procedure with sequential use of Liraglutide at 6 months compared to those receiving Liraglutide and then undergoing the POSE 2.0 procedure at 6 months.

DETAILED DESCRIPTION:
The growing impact of obesity worldwide has consequences on patients' quality of life, numerous weight-related comorbidities, and global economic costs. Numerous therapies for obesity treatment involve lifestyle modifications, pharmacotherapy, and procedural intervention, though many limitations exist. Bariatric surgery has been shown to be the most durable and effective; however, the invasive nature and complications, such as micronutrient deficiencies, often damper enthusiasm for these procedures. Furthermore, it is often unavailable to those with class I or II obesity. Two emerging modalities have shown promising results for sustained weight loss: minimally invasive endoscopic bariatric therapies such as the POSE2.0 procedure and GLP-1 agonists, including Liraglutide. Recent data examining these methods individually have demonstrated weight loss of 5-10% percent total body weight for Liraglutide vs. 15-20% for POSE2.0. No studies have evaluated these therapies head-to-head and in combination. This pilot randomized crossover trial aims to investigate the weight loss outcomes between Liraglutide and POSE2.0 procedure. The investigators will recruit 25 subjects in each of the two intervention groups for a 6-month treatment period with each therapy. At 6 months, if the subject has not attained a BMI less than or equal to 30 kg/m2 in the Liraglutide arm or 28 kg/m2 in the POSE2.0 arm, they will cross over to the other intervention to utilize the combination of POSE2.0 and Liraglutide for additional 6 months. As per clinical guidelines, The cross-over criteria are congruent with accepted clinical guidelines for the use of these interventions. If the patient does not achieve greater than 5% total body weight loss on Lirglutide alone by 3 months as per accepted clinical criteria, the Liraglutide will not be continued as per clinical recommendation and the subject will cross over to the POSE2.0 procedure at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adult patients (22 years of age or above and less than 60 years of age)
* Body mass index (BMI) ≥30 and <40 kg/m2
* Provision of signed and dated informed consent form.
* Subject agrees to be compliant with study requirements and adhere to dietary & exercise recommendations for the duration of the study.
* If female, be either post-menopausal, surgically sterile, or agree to practice birth control during year of study and have negative serum HCG at screening/baseline.
* Absence of current severe systemic disease (including, but not limited to: coronary artery disease, chronic obstructive pulmonary disease, congestive heart failure, cancer, and chronic renal disease).
* Agrees not to undergo any additional weight loss interventional procedures or liposuction for 12 months following study enrollment.
* Have not taken any prescription or over the counterweight loss medications OR those that can suppress appetite/induce weight loss for at least 6 months and agrees not to utilize for 12 months following study enrollment (including all stimulant medication).
* Subjects must be willing to possibly forego any future weight loss procedures (i.e. Vertical Sleeve Gastrectomy) following the study given the unknown long-term effects.
* Residing within a reasonable distance from the Investigator's treating office (~50 miles) and willing and able to travel to the Investigator's office to complete all routine follow-up visits

Exclusion Criteria:

* Prior bariatric, gastric or esophageal surgery.
* Esophageal stricture or other anatomy and/or condition that could preclude passage of endoluminal instruments or procedure execution.
* Moderate gastro-esophageal reflux disease (GERD), defined as symptoms that cause subject severe discomfort, compromise performance of daily activities, and/or condition is not entirely controlled with drug therapy.
* Large hiatal hernia (>3 cm) by history or as determined by pre-enrollment endoscopy.
* Pancreatic insufficiency/disease.
* History of gastroparesis or symptoms that would be suggestive of gastroparesis or generalized dysmotility (e.g. esophago-gastric motility issues and lower esophageal sphincter abnormalities).
* Pregnancy or plans of pregnancy in the next 12 months.
* History of a known diagnosis or pre-existing symptom of rheumatoid arthritis, scleroderma, system lupus, or other autoimmune connective tissue disorder.
* Immunosuppressive medications or systemic steroids (i.e., oral prednisone) within 6 months of Visit 1. Intranasal/inhaled steroids are acceptable.
* Unable or unwilling to avoid use of aspirin and/or non-steroidal anti-inflammatory drugs (NSAIDs), or other medications known to be gastric irritants beginning two weeks prior to enrollment and throughout the entire study.
* History of inflammatory disease of the GI tract; coagulation disorders; hepatic insufficiency or cirrhosis.
* Active gastric erosion, lesion, or gastric/duodenal ulcer.
* History of or current platelet or coagulation dysfunction, such as hemophilia.
* History or present use of insulin or insulin derivatives for treatment of diabetes.
* Type II Diabetes Mellitus (as defined by HgbA1c >6.5%) for greater than 11 years at the time of enrollment.
* If smoker, plans to quit smoking in the year after enrollment.
* Portal hypertension and/or varices.
* Patient has a history of drug or alcohol abuse or positive at screening for drugs of abuse. - Patient is currently using marijuana/cannabis for either medicinal or recreational use, or has plans to start using over the next 12 months.
* Present or history of psychosis, bipolar disease, or obsessive-compulsive disorder after pre-enrollment history and medical /psychological assessment.
* Uncontrolled depression after pre-enrollment psychological and medical assessment.
* If significant findings for depression and/or suicidal ideation are identified, the psychologist(s) assigned to the study will be contacted and arrangement will be made for immediate intervention according to the Institution's standard procedure.
* Non-ambulatory or has significant impairment of mobility (i.e. cannot ambulate for 30 minutes).
* Known hormonal or genetic cause for obesity including untreated hypothyroidism (TSH >5.0 U/ml).
* Participating in another clinical study.
* Subjects with a personal history of allergic/anaphylactic reactions including hypersensitivity to the drugs or materials that will be utilized in the study procedure.
* Physician's assessment that the subject is not an appropriate candidate.
* Breastfeeding
* Personal or family history of medullary thyroid cancer or MEN2
* Suicidal ideation and behavior.
* Injection site reaction

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2025-01-03 (Estimated); Study Completion 2026-01-03 (Estimated)

PRIMARY OUTCOMES:
Mean percent total body weight loss at 6 months in each arm of the study | 6 months
  Percent total body weight loss
Percentage of subjects with ≥5 percent total body weight loss at 6 months in each arm at 6 months | 6 months
  Percentage of subjects with ≥5 percent total body weight loss
The incidence, frequency, and severity of adverse events related to treatment with the device and procedure as well as medication will be reported. | at 6 months
  Adverse events

SECONDARY OUTCOMES:
Mean percent TBWL in each arm of the study at 12 months. | 12 months
  Mean percent total body weight loss in each arm at 12 months.
Percentage of subjects with ≥10 percent TBWL at 6 months in each arm. | 6 months
  Percentage of subjects with ≥10 percent TBWL at 6 months.
Percentage of subjects with ≥10 percent TBWL at 12 months in each arm. | 12 months
  Percentage of subjects with ≥10 percent TBWL at 12 months in each arm.
Change from baseline of the Controlled Attenuation Parameter (CAP) dB/m measured by Fibroscan at 6 months in each arm | 6 months
  Controlled Attenuation Parameter (CAP) each arm (dB/m)
Change from baseline of the Controlled Attenuation Parameter (CAP) dB/m measured by Fibroscan at 12 months in each arm. | 12 months
  Controlled Attenuation Parameter (CAP) each arm (dB/m)

OTHER OUTCOMES:
Change from baseline of liver fibrosis score (kilopascal) measured by Fibroscan at 12 months. | 12 months
  liver fibrosis score (kilopascal)

CONTACTS AND LOCATIONS:
Overall Officials: Maryam AlKhatry, MD, Principal Investigator — EHS
Locations (1):
- Ibrahim Bin Hamad Obaidullah Hospital, Ras al-Khaimah, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No